CLINICAL TRIAL: NCT04713514
Title: Randomized Phase II Study Comparing Neo-epitope Based Vaccine OSE2101 (TEDOPI®) With or Without Anti-PD1 (Pembrolizumab) Versus Best Supportive Care as Maintenance Treatment in Platinum-sensitive Recurrent Ovarian Cancer Patient With Controlled Disease After Platinum-based Chemotherapy
Brief Title: OSE2101 Alone or in Combination With Pembrolizumab vs BSC in Patient With Platinum-sensitive Recurrent OC
Acronym: TEDOVA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: OSE Immunotherapeutics (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-OV244b; 2020-004364-25 (EudraCT Number); ENGOT-ov58 (Other: ENGOT)
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Platinum-sensitive Ovarian Cancer; Relapsed Ovarian Cancer
Keywords: Maintenance therapy; Immunotherapy; Cancer vaccine; Cold tumor; Relapse; Pembrolizumab; TEDOPI
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A : Best Supportive Care (No Intervention): Observational arm (Standard of care)
- Arm B : OSE2101 (Experimental): OSE2101 monotherapy - subcutaneous injection on day 1, every 3 weeks for 7 doses then every 6 weeks up to week 48 and then every 12 weeks until intolerance, disease progression, or up to 2 years.
  OSE2101 vaccine is an emulsion of peptides suspension in in Montanide® ISA 51 adjuvant and containing 0.5 mg/mL of each 10 synthetically manufactured peptides (5.0 mg/mL total peptide) in 1.5 mL of emulsion.
  Interventions: Drug: OSE2101
- Arm C : OSE2101 + Pembrolizumab (Experimental): OSE2101 (subcutaneous injection on day 1, every 3 weeks for 7 doses then every 6 weeks up to week 48 and then every 12 weeks until intolerance, disease progression, or up to 2 years) + pembrolizumab (400 mg IV infusion on day 1 every 6 weeks until intolerance, disease progression, or up to 2 years.
  Interventions: Drug: OSE2101; Drug: Pembrolizumab 25 MG/ML [Keytruda]

INTERVENTIONS:
Drug: OSE2101 — subcutaneous injection on day 1, every 3 weeks for 7 doses then every 6 weeks up to week 48 and then every 12 weeks until intolerance, disease progression, or up to 2 years.
  Other Names: TEDOPI®
  Arms: Arm B : OSE2101; Arm C : OSE2101 + Pembrolizumab
Drug: Pembrolizumab 25 MG/ML [Keytruda] — 400 mg IV infusion on day 1 every 6 weeks until intolerance, disease progression, or up to 2 years.
  Other Names: KEYTRUDA®; MK-3475
  Arms: Arm C : OSE2101 + Pembrolizumab

SUMMARY:
The proposed study is an international randomized phase II, multicenter, open-label, three arms trial to assess best supportive care (BSC) vs OSE2101 and vs OSE2101 + pembrolizumab as maintenance treatment for patients with platinum sensitive relapsed ovarian cancers, previously treated with chemotherapy (regardless of the number of prior lines of platinum-based chemotherapy), bevacizumab (if eligible) and a PARP inhibitor (if eligible).

Patients in Complete Response, Partial Response, or Stable Disease at the end of chemotherapy with at least 4 cycles of platinum based chemotherapy will be randomized in one of the three arms (randomization 1:1:2). They will receive one or the two study treatments or BSC until progression, or intolerance, or up to 2 years (from 1st study treatment dose).

DETAILED DESCRIPTION:
The only therapeutic option for ovarian cancer patients presenting platinum sensitive relapse post- both bevacizumab and a PARPi is a platinum combination x 6 cycles followed by observation. There is no currently approved maintenance therapy in this setting. There is an urgent need for novel strategies for OC in relapse post bevacizumab and PARPi, in particular for novel maintenance strategies to prolong chemotherapy-free intervals.

One attractive strategy to turn OC from 'cold' tumors into a 'hot' tumor is via vaccination with tumor associated, or specific epitopes that have been modified to increase MHC and TCR binding.

OSE2101 is a multi-neoepitope vaccine covering relevant TAAs in OC, including p53 (mutated in 95% of high-grade OC). In addition, the combination of OSE2101with an ICI may most effectively harness anti-tumor immunity.

If novel IO approaches are proposed in OC, they should be investigated early in the disease setting when host immunity is still robust, and with low tumor burden (platinum sensitive relapse and after 6 cycles of platinum chemotherapy).

The hypothesis being tested is that OSE2101 alone or in combination with Pembrolizumab as maintenance treatment in patients with ovarian cancer platinum-sensitive relapse could potentially bring benefit to subjects with high unmet medical need.

A total of 180 patients with HLA-A2 positive phenotype will be randomized using an Interactive Web Response System (IWRS) according to the following stratification factor:

• Best response to platinum therapy: SD vs PR/CR

In a 1:1:2 ration on the 3 study arms:

* Arm A (n=45): Observation/best supportive care
* Arm B (n=45): OSE2101: every 3 weeks until week 18, then every 6 weeks up to week 48, then every 12 weeks until disease progression, intolerance, patient withdrawal of consent or up to 2 years
* Arm C (n=90): OSE2101 + Pembrolizumab: OSE2101 same schedule as arm B plus pembrolizumab IV every 6 weeks until disease progression, intolerance, patient withdrawal of consent or up to 2 years

Patient with phenotype HLA-A2 negative will be followed in a separate cohort to record treatment and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent document for the study, willing and able to comply with protocol requirements, including:

   1. HLA-A2 phenotype determination by genetic test (blood)
   2. participation in translational research in HLA-A2 positive
   3. authorization for long term follow up if HLA-A2 negative
2. Histologically proven non-mucinous epithelial ovarian cancer
3. Positive HLA-A2 phenotype
4. Age ≥ 18 years
5. ECOG Performance Status (PS) 0-1
6. Clinical or radiological relapse of a platinum sensitive ovarian cancer regardless of the number of prior lines of platinum-based chemotherapy, as long as each prior line fulfilled the platinum sensitive criteria defined as complete response, partial response or stable disease according to RECIST 1.1 at the end of a platinum-based chemotherapy. Patient must have received at least 4 infusions of platinum during the last line of platinum-based chemotherapy
7. Previously treated with a PARP inhibitor or not eligible to PARPi (i.e ineligibility due to not complete or partial response to chemotherapy)
8. Prior therapy with bevacizumab or with contra-indication to bevacizumab (i.e arterial thromboembolic events, history of intestinal perforation, any other contra-indications according to the SmPC)
9. Patient may have received prior immune checkpoint inhibitor (ICI), such as anti-PD-(L)1 or anti-CTLA-4 antibody and had a relapse after receiving the ICI without concomitant chemotherapy for at least 6 months (as treatment or maintenance)
10. Randomization must be within 8 weeks of last dose of chemotherapy
11. Adequate organ function Adequate marrow function White blood cell (WBC) ≥ 3000/ mm3 Neutrophils ≥ 1500/ mm3 Platelets ≥ 100 × 103/mm3 (in the absence of transfusion within 2 weeks from before randomization) Haemoglobin ≥ 9 g/dL (in the absence of transfusion within 2 weeks from before randomization) Adequate other organ functions ALT and AST ≤ 2.5 × ULN, unless liver metastases are presents in which case they must be ≤ 5.0 × ULN Total bilirubin ≤ 1.5× ULN (except Gilbert Syndrome: < 3.0 mg/dL)

    Serum creatinine ≤ 1.5 × ULN or creatinine clearance (CrCl) ≥ 40 mL/min (measured using the Cockcroft-Gault formula below):

    Female CrCl = (140 - age in years) × weight in kg × 0.85 72 × serum creatinine in mg/dL
12. Archival or fresh (if possible) tumor tissue must be available for evaluating relevant biomarkers.
13. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to treatment allocation, and have to use of highly effective contraception during the treatment period and for at least 180 days after the last dose of study treatment
14. Stated willingness to comply with all study procedures and availability for the duration of the study
15. For countries where this will apply to : a subject will be eligible for randomization in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

1. Patient with contra-indications to immune therapies
2. Ongoing immunotherapy (checkpoint inhibition, antigen immunotherapy that would be scheduled to continue concomitantly to the study)
3. Use of any of the following immunomodulatory agents within 30 days prior to the first dose of study drug: Systemic corticosteroids (at dose higher than 10 mg/day equivalent prednisone); if systemic corticoid use, corticoid must be stopped at least 7 days before study treatment start Interferons Interleukins Live vaccine

   Note: Examples of live vaccines include, but are not limited to, the following:

   measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed as other killed vaccines, if done at least 2 weeks prior the first dose of study drug; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
4. Prior cancer vaccine therapy
5. Patient eligible for cytoreductive surgery at the time of inclusion
6. Patient with clinical, radiological or biological progression (according GCIG criteria) at the end of last chemotherapy
7. Prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.

   A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
8. Patient with active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
9. History of serious adverse reactions, including anaphylaxis and related symptoms such as hives and respiratory difficulty following administration of any vaccines, or a history of hypersensitivity, specifically to any components of study vaccine
10. Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or other in situ cancer considered as cured) unless the patient has been free of the disease for at least 5 years.
11. Immune-deficient status (patients with HIV, immunosuppressive treatment, haematological malignancies, and previous organ transplantation)
12. History of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease that requires steroids.
13. History of any chronic hepatitis as evidenced by:

    Positive test for hepatitis B surface antigen Positive test for qualitative hepatitis C viral load (by polymerase chain reaction [PCR]) Note: Subjects with positive hepatitis C antibody and negative quantitative hepatitis C by PCR are eligible. History of resolved hepatitis A virus infection is not an exclusion criterion
14. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following: Myocardial infarction or stroke/transient ischemic attack within the past 6 months Uncontrolled angina within the past 3 months History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III-IV, pericarditis, significant pericardial effusion, or myocarditis) Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes) QT interval corrected for heart rate using Fridericia's formula (QTcF) prolongation > 480 msec Cardiovascular disease-related requirement for daily supplemental oxygen therapy
15. Subjects with known or suspected CNS metastases, untreated CNS metastases, are excluded. However, subjects with controlled brain metastases will be allowed to enroll. Controlled brain metastases are defined as no radiographic progression for at least 4 weeks following radiation and/or surgical treatment (or 4 weeks of observation if no intervention is clinically indicated), and off of steroids for at least 2 weeks, and no new or progressive neurological signs and symptoms.
16. Any major surgery within 4 weeks of study drug administration. Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before date of randomization.
17. Patients who has severe hypersensitivity (Grade 3 or higher) to pembrolizumab and/or any of its excipients (refer to the IB for a list of excipients).
18. Patients who has an active infection requiring systemic therapy.
19. Any acute medical condition that in the opinion of the investigator may obscure the ability to observe the safety or activity of the study vaccine treatment
20. Any mental or psychiatric condition that, in the opinion of the investigator, is likely to compromise the ability to adhere to the protocol schedule
21. Life expectancy of less than 12 weeks
22. Pregnant or breastfeeding women
23. Concurrent participation in any other investigational study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from date to randomization to date of event, assessed up to 4 years
  Progression-free survival (PFS) is the time from randomization to progression measured radiologically using RECIST v1.1 guidelines as reported by the investigator or death, whatever the cause, whichever comes first. Patients alive and free of progression at the cut-off date will be censored at the last tumor assessment date

SECONDARY OUTCOMES:
Objective response rate (ORR) | from date to randomization to date of event, assessed up to 4 years
  Objective response rate is defined using RECIST v1.1. Best overall response is defined as the best radiological response observed over the whole evaluation period before progression or subsequent anti-cancer treatment. Proportion of partial and complete responses over the treated population will be computed.
Incidence of treatment emergent adverse events | from date to randomization to date of study end, assessed up to 4 years
  Incidence of treatment emergent adverse events will be assessed based on NCI CTC-AE version 5.0 grade and according MedDRA terms (version 23.0)
Time to subsequent first treatments (TTST-1) | from date to randomization to date of event, assessed up to 4 years
  Time to subsequent treatment (TTST) is the time from randomization to initiation of a first subsequent treatment (including treatment change due to toxicity or investigator's decision). Deaths will be counted as events. Patients alive and not receiving a subsequent treatment will be censored at the last assessment date.
Time to subsequent second treatments (TTST-2) | from date to randomization to date of event, assessed up to 4 years
  Time to subsequent treatment (TTST) is the time from randomization to initiation of second subsequent treatment (including treatment change due to toxicity or investigator's decision). Deaths will be counted as events. Patients alive and not receiving a subsequent treatment will be censored at the last assessment date.
Overall Survival (OS) | from date to randomization to death from any cause, assessed up to 4 years
  Overall Survival (OS) is defined as time from randomization to the date of death, whatever the cause. Patients alive at the cut-of date will be censored at the last date they are known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra LEARY, MD,PHD, Principal Investigator — GINECO - Gustave Roussy
Locations (40):
- Belgium (3):
  - UZ Leuven, Leuven
  - Centre Hospitalier de l'Ardenne Vivalia, Libramont
  - Centre Hospitalier Universitaire de Liège, Liège
- France (31):
  - ICO Paul Papin, Angers
  - Institut du Cancer Avignon-Provence, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre d'Oncologie et de Radiothérapie 37, Chambray-lès-Tours
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean PERRIN, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - CHU Grenoble-Alpes - Site Nord (La Tronche), Grenoble
  - Centre Oscar Lambret, Lille
  - CHU Limoges - Dupuytren, Limoges
  - Hôpital Privé Jean Mermoz, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM - Val d'Aurelle, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Hôpital Pitié-Salpêtrière - AP-HP, Paris
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Diaconesses-Croix Saint-Simon, Paris
  - Center Hospitalier de Pau, Pau
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - Centre Eugène Marquis, Rennes
  - ICO - Centre René Gauducheau, Saint-Herblain
  - CHU de Saint-Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - Centre Hospitalier Broussais, St-Malo
  - Institut de Cancérologie de Strasbourg Europe - ICANS, Strasbourg
  - Institut Claudius Régaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (6):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Evang. Kliniken Essen-Mitte GmbH, Essen
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Universitätsmedizin Mannheim GmbH, Mannheim
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Derived] Kabirian R, Tredan O, Marme F, Paoletti X, Eberst L, Lebreton C, De La Motte Rouge T, Sabatier R, Angelergues A, Fabbro M, Van Gorp T, Mansi L, Gladieff L, Kaczmarek E, Alexandre J, Grellety T, Favier L, Welz J, Frenel JS, Leary A. TEDOVA: vaccine OSE2101 +/- pembrolizumab as maintenance in platinum-sensitive recurrent ovarian cancer. Future Oncol. 2024;20(35):2699-2708. doi: 10.1080/14796694.2024.2386922. Epub 2024 Aug 19. PMID 39155847